CLINICAL TRIAL: NCT02198989
Title: Effects of Peer Support and Yoga Music on T2DM With Depression and Sleep Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang Ning (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor-Investigator, Guang Ning, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCEMD-022
Record Dates: First submitted 2014-07-10; First posted 2014-07-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- peer support and yoga music therapy (Experimental): Patients in the group will receive peer support and yoga music therapy before bed.
  Patients in the group will received the group education courses and clinical medical therapy.
  Interventions: Behavioral: peer support and yoga music therapy
- Control group (No Intervention): Patients in the group will received the group education courses and clinical medical therapy.

INTERVENTIONS:
Behavioral: peer support and yoga music therapy — Patients in the intervention group will receive peer support and yoga music therapy before bed.
  Arms: peer support and yoga music therapy

SUMMARY:
40 patients with Type 2 Diabetes Mellitus who also have sleep disorders and mild depression in the community will be recruited and stochastically divided into the intervention group and the control group. Both groups will take the same group education courses including DSME (Diabetes Self-management Education), psychological support, improvement in sleep. Patients in the intervention group will receive peer support and yoga music therapy before bed. The observation period will last for 6 months so as to evaluate the benefits of peer support and yoga music therapy in sleep quality improvement and glycemic control of type 2 diabetic patients with sleep disorders and mild depression.

DETAILED DESCRIPTION:
Research Method:

This study is an open- label controlled randomized cluster trial with the sample size estimated by the improvement of Pittsburgh Sleep Quality Index（PSQI） score. 40 eligible and voluntary Type 2 diabetic patients will be recruited among the patients with health records in the community. Baseline assessment such as demography, sleep quality, depression, physical exam and biochemical index will be performed on the patients who will have signed the informed consents.

The study will use the method of randomized to classify the enrolled units into 2 groups, each group has 20 people. Both groups will receive regular diabetes medication and group education courses including Diabetes Self-management Education(DSME), psychological support, improvement in sleep. The intervention group will be under the guidance of two well-trained peer supporters to carry out group activities. Each supporter will be in charge of 10-15 patients. Starting with peer support therapy in the first three months, the intervention group will then take Yoga music therapy before bed for another three months and be given support and guidance by the peer supporters.

Compare the baselines and variations of two group's sleep, depression, blood sugar and related biochemical indicators, and self-management, life quality, medication and other aspects at the third month and sixth month. The final evaluation will show the effect and related influencing factors of peer support and yoga music therapy in helping Type 2 diabetic patients who have sleep disorders and mild depression to improve their sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed type 2 diabetes patients (ICD9) according to the medical record and patient's disease history
* Diagnosis type 2 diabetes more than 6 months
* 40 Years to 84 Years old
* Sleep-disordered patients (PSQI scores≥7)
* Mild depression condition（14 ≥PHQ-9 scores≥ 5 分）
* Have a stable T2DM condition，without any other diseases affect patients' sleep
* Agree to participate in the study and have signed the Inform Consent Form

Exclusion Criteria:

* Terminal illnes
* Hearing loss or severe visual disorder
* Life expectancy is less than 12 months
* Primary sleep apnoea syndrome
* Serious physical pain that affect the quality of sleep
* Using drugs that affect the quality of sleep
* Individuals with histories of Alcohol or Drug Abuse
* Patients with high risk for sleep apnea syndrome(STOP scores ≥3 )
* Planned to receive selective surgery within 3months
* Observed mental confusion suggesting dementia
* Ongoing psychiatric care
* Paralysis or residence in a long-term care facility

Ages: 40 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Score on Pittsburgh Sleep Quality Index（PSQI） | 9 months
Score on Patient Health Questionnaire (PHQ-9) | 9 month
HbA1c | 9 months

SECONDARY OUTCOMES:
BMI | 9 months
Insulin resistance measured as HOMA-IR | 9 months
  HOMA-IR = (FINS×FPG) / 22.5

CONTACTS AND LOCATIONS:
Overall Officials: Liebin Zhao, MSM, Study Chair — Center of Diabetes, Ruijin Hospital, Shanghai Jiao Tong University of Medicine
Locations (1):
- Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China